CLINICAL TRIAL: NCT01002118
Title: Feasibility of Omega-3 Fatty Acid Supplementation in Adult Hemodialysis Patients
Brief Title: Feasibility Study of Omega-3 Fatty Acids in Dialysis Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit eligible subjects; no data analyzed
Sponsor: University of Iowa (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Jennifer G. Robinson, Principal Investigator, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200801761
Record Dates: First submitted 2009-10-23; First posted 2009-10-27 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Cardiovascular Disease
Keywords: heart rate variability; Dialysis
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Omacor

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 4 capsules inert oil Placebo each day for 16 weeks
  Interventions: Drug: Placebo
- Omega-3 Fatty Acid Ethyl Esters (Active Comparator): 4 capsules Omega-3 Fatty Acid Esters each day for 16 weeks
  Interventions: Drug: Omega-3 Acid Ethyl Esters

INTERVENTIONS:
Drug: Omega-3 Acid Ethyl Esters — 1 gram capsules Omega-3 Acid Ethyl Esters for a total of 4 grams (4 capsules) per day for 16 weeks
  Other Names: Lovaza Omega-3 Acid Ethyl Esters 4g capsule
  Arms: Omega-3 Fatty Acid Ethyl Esters
Drug: Placebo — 4 capsules each day for 16 weeks
  Arms: Placebo

SUMMARY:
Cardiovascular disease and mortality is the largest comorbidity within the dialysis population. Nearly 50% of hemodialysis patients will have congestive heart failure at initiation. According to the most recent United States Renal Data System (USRDS), 40% of incident dialysis patients will have a cardiovascular event or die within the first 9 months of dialysis. It has been postulated that Omega-3 fatty acids could provide beneficial cardioprotection in hemodialysis patients. The investigators propose to evaluate Omega-3 fatty acid doses on cardiovascular parameters in an incident hemodialysis population. Initially, this will be a pilot study. Ultimately, the information will be used to adequately plan for a larger intervention trial using Omega-3 fatty acids in incident hemodialysis patients.

DETAILED DESCRIPTION:
Cardiovascular disease and mortality is the largest comorbidity within the dialysis population.

Nearly 50% of hemodialysis patients will have congestive heart failure at initiation. According to the most recent USRDS data, 40% of incident dialysis patients will have a cardiovascular event or die within the first 9 months of dialysis. The risk of sudden cardiac death is estimated to be 6.9% per year of dialysis. Despite this, a recent study found that only 8% of dialysis patients received an implantable defibrillator. Numerous studies have looked at the acute cardiac effects of hemodialysis. Changes in the QT interval, elevations in troponins, increased heart rate variability and heart have all been noted. The mechanisms behind these changes and potential preventative measures remain unknown. It has been postulated that Omega-3 fatty acids could provide beneficial cardioprotection in hemodialysis patients. In nonhemodialysis populations, omega-3 fatty acids (FA) have established anti-arrhythmic properties and have been shown to reduce the risk of sudden death and to reduce cardiac mortality. In a study of hemodialysis patients, a high dose of omega-3 FA (5 grams daily) had beneficial effects on electrocardiographic (ECG) surrogate markers of sudden death, such as heart rate, heart rate variability, and baroreflex sensitivity. One small 2-year study of 1.7 grams omega-3 FA in 206 hemodialysis subjects showed a significant reduction in myocardial infarction but was not large enough to detect an effect on cardiac or total mortality. While these studies are suggestive, the potential therapeutic benefit remains unclear and the appropriate dose of Omega-3 in dialysis patients to achieve benefit is unknown. Doses of Omega-3 that have shown electrocardiogram benefits were high and require 6-8 capsules daily. Long-term adherence is likely to be suboptimal with this high pill burden. Studies with smaller doses have been of insufficient size to determine any cardiovascular benefit. We propose to evaluate two Omega-3 fatty acid doses on cardiovascular parameters in a hemodialysis population. Initially, this will be a pilot study. Ultimately, the information will be used to adequately plan for a larger intervention trial using Omega-3 fatty acids in incident hemodialysis patients. I.5 Specify your research question(s), study aims or hypotheses (do not indicate "see protocol") Specific aim 1. Determine recruitment and medication adherence rates Recruitment will take place over 6 months and include incident hemodialysis patients with a 4 month follow-up. Total expected time for the pilot is one year. Participants will be randomized to either moderate dose Omega-3 (4 grams), or 4 tables of placebo. Rates of participation, medication adherence and drop out rates will be used to plan future trials. HawkIRB https://hawkirb.research.uiowa.edu/hawkirb/summary/projects.page?mode=pf&OID=5961841[1/27/2010 2:46:08 PM] Specific aim 2. Assess the effectiveness of two Omega-3 fatty acid doses compared to placebo on electrocardiographic parameters. All participants will have a cardiovascular evaluation at baseline and at end of study. This will include a 48-hour Holter monitor, vital signs and blood studies of various cardiovascular risk markers. Specifically, we will be assessing heart rate variability, heart rate and QT dispersion.

Specific aim 3. Assess the side effect profiles of 3.4 g Omega-3 fatty acids to placebo.

The success of future trials will require subject compliance with therapy. By evaluating the side effects of Omega-3, we will be better able to determine the tolerability for future studies.

I Selection of study endpoints. Since this is a feasibility study there will be insufficient power to detect changes in physiologic parameters. Omega-3 FA have been shown to beneficially influence autonomic function parameters measured by 48-hour Holter we have selected as our secondary endpoints changes HRV, heart rate, and QT duration for a dose-ranging study. Blood samples will be obtained and properly stored for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Initiated dialysis in past 3 months
* Signed informed consent
* Attending University of Iowa dialysis unit for duration of the study

Exclusion Criteria:

* Age >70
* Unable to provide consent
* Currently taking fish oil supplementation
* rhythm other than sinus
* implantable cardioverter-defibrillator
* pacemaker
* myocardial infarction,revascularization or unstable angina in past 3 months
* other hospitalization in past 3 months
* symptomatic heart failure
* known left ventricular ejection fraction < 30%
* history of a significant bleeding disorder
* severe bleeding episode requiring hospitalization in past 3 months (GI bleed or hemorrhagic stroke)
* unexplained HgB drop > 2 gm/dl in past 3 months
* chronic warfarin or anti-coagulation therapy (such as Lovenox)
* pregnant or nursing mothers
* allergic to fish, fish oil or fish products
* Participation in other trials of investigational products
* other characteristics as determined by the investigator that would make sudy participation inappropriate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-01-25 (Actual); Primary Completion 2011-02-23 (Actual); Study Completion 2011-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Robinson, MD MPH, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Omega-3 Fatty Acid: Omega-3 Acid Ethyl Esters: 1 gram capsules for a total of 4 grams (4 capsules) per day for 16 weeks
Period: Overall Study
Arm/Group | Omega-3 Fatty Acid
Started | 1
Randomized Only Patient | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Omega-3 Fatty Acid
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Holter monitor [Count of Participants; unit: Participants] | 1

OUTCOME MEASURES:

1. Primary Outcome: Determine Recruitment Rates
Description: Determine recruitment by number eligible/number enrolled
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Omega-3 Fatty Acid
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: Assess the Effectiveness of Omega-3 Fatty Acid Compared to Placebo on Electrocardiographic Parameters.
Description: percent of subjects with significant arrhythmia present on Holter electrocardiography
Time Frame: 4 months
Measure: Number; unit: percentage of Holter montiors obtained
Arm/Group | Omega-3 Fatty Acid
Number analyzed (Participants) | 1
percentage of Holter montiors obtained | 0

3. Secondary Outcome: Medication Adherence
Description: percent of pills taken each month calculated as number of pills taken/number of pills dispensed
Time Frame: 4 months
Measure: Number; unit: percentage of pills
Arm/Group | Omega-3 Fatty Acid
Number analyzed (Participants) | 1
percentage of pills | 100

ADVERSE EVENTS:
Arm/Group | Omega-3 Fatty Acid
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No